CLINICAL TRIAL: NCT04769973
Title: The PD Life Study: Exploring the Treatment Burden and Capacity of People With Parkinson's and Caregivers
Brief Title: Treatment Burden in Parkinson's
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: Southern Health NHS Foundation Trust (Other); Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 62623; 277464 (Other: IRAS)
Record Dates: First submitted 2021-01-15; First posted 2021-02-25 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease; Parkinson
Keywords: Treatment Burden; Burden of Treatment
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Work Packages 1 - 3: Work Package 1: Interviews with 15-20 people with Parkinson's and 15-20 caregivers.
  Work Package 2: National Survey with up to 2000 participants
  Work Package 3: Two to four Focus Groups with key stakeholders (6-10 participants per focus group)

SUMMARY:
Background:

People with Parkinson's (PwP) have many symptoms including tremor, stiffness, slow movements, constipation, urinary incontinence and mental health issues. They are often older and have other long-term health conditions. PwP need to do many things to look after their health including manage multiple medications, attend healthcare appointments and lifestyle changes such as improving diet and exercise.

The effort of looking after their health and its impact on them is termed 'treatment burden'. Some PwP need help from their family or friends (caregiver) to complete these tasks. Caregivers may also experience treatment burden themselves when caring for someone with Parkinson's. People's ability to manage treatment burden is termed 'capacity' and is influenced by physical, mental, social and economic factors. People are overburdened when the workload of looking after their health exceeds their capacity. This can lead to poor adherence with treatment, poor quality of life and worse health outcomes.

Aim:

To understand the factors that influence treatment burden and capacity in PwP and caregivers of PwP.

Methods:

Interviews with PwP and caregivers will identify factors that influence treatment burden and capacity. These factors will be explored further in a national survey for PwP and caregivers through Parkinson's UK. The investigators will form focus groups with PwP, caregivers, voluntary sector representatives, healthcare professionals, policy makers and managers through Parkinson's Excellence Networks to discuss and prioritise recommendations for change.

Outcomes:

The investigators will disseminate recommendations of ways to reduce treatment burden and improve future experiences of PwP and caregivers.

DETAILED DESCRIPTION:
This is a mixed-methods study that will be conducted over three work packages as described below and will be completed in 24 months. The investigators will have patient and public involvement throughout the study.

Work Package 1 - Interviews:

The investigators will interview 15-20 PwP and 15-20 caregivers (face-to-face, telephone or video calls) recruited from Parkinson's clinics in Hampshire and Dorset to identify factors that influence treatment burden and capacity among PwP and caregivers of PwP. Participants will be eligible to take part in the study if they have a diagnosis of Parkinson's or is a caregiver for someone with Parkinson's, and able to give informed consent. The investigators will use purposive sampling to include both genders, a range of ages, severity of Parkinson's and caregiver relationships. Potential eligible participants will be identified by the clinical team. Written consent will be obtained prior to each interview. Interviews will be audio-recorded and transcribed. The investigators will take an inductive approach to identify emerging themes until no new information arises.

Work Package 2 - National Survey:

Results from the interviews will then inform the development of a national survey for PwP and caregivers. The national survey will for the first time quantify treatment burden using the Multimorbidity Treatment Burden Questionnaire (MTBQ) and capture aspects of capacity such as severity and duration of Parkinson's, social and economic resources, medications, frailty and health literacy. Participants with mild, moderate and severe Parkinson's will be recruited with agreed support from Parkinson's UK and from Parkinson's clinics. Participants will be eligible to take part in the study if they have a diagnosis of Parkinson's or is a caregiver for someone with Parkinson's, and able to give informed consent. Each participant will be able to complete a separate survey online or on paper.

The investigators will collect the following data from participants:

1. Sociodemographic data: age, sex, ethnicity, cohabitation status, living situation, presence of caregiver, employment status, education level, access and ability to drive, access to information technology
2. Multimorbidity Treatment Burden Questionnaire (MTBQ
3. Information about Parkinson's including: - i) Year of diagnosis ii) Self-reported Parkinson's severity (Hoehn and Yahr)
4. Other health conditions
5. Single-item health literacy score
6. Medications use and frequency
7. Healthcare use of the person with Parkinson's in the last 12 months e.g. primary, secondary and urgent care
8. Assessment of frailty with PRISMA-7: a brief 7-item self-reported questionnaire
9. Quality of Life Measures with the 12-item Short Form Health Survey (SF-12v2)
10. A single question to consider the overall effort of looking after health

The investigators will also collect data regarding non-motor symptoms from PwP using the Parkinson's Disease Non-Motor Symptoms Questionnaire.

The investigators will collect the following data from caregivers of PwP: -

1. Information about the Parkinson's of the person they care for including: - i) Issues with memory, mood and hallucinations ii) Awareness of deterioration from the person with Parkinson's
2. Zarit Burden Interview: a 12-item scale that assesses the caregiver burden.

Work Package 3 - Focus groups and Dissemination:

Working with Wessex Parkinson's Excellence Network, the investigators will hold two to four focus groups with key stakeholders including PwP, caregivers, voluntary sector representatives, healthcare professionals, policy makers and managers. Participants will be recruited from each local area (Hampshire and Dorset) through Parkinson's clinics, support groups and local services depending on the findings from the interviews and surveys. Each focus group will have 6-10 participants and will be moderated by a member of the research team. Written consent will be obtained from each participant prior to the focus group. Focus groups will be conducted either face-to-face at a neutral location or conducted via video call. Each focus groups will be audio-recorded using a digital recorder with consent and transcribed for further data analysis. The focus groups will discuss the overall study findings and aim to develop and prioritise recommendations of ways to reduce treatment burden and enhance capacity among PwP and their caregivers.

The investigators will then hold a dissemination event to share the outcomes with people affected by Parkinson's with support from Parkinson's UK and the Academic Health Science Networks. The investigators will work closely with Parkinson's UK Excellence Networks to share knowledge and implement changes that improve treatment burden and enhance capacity among PwP and caregivers. The findings will be disseminated through publications in peer-reviewed journals and presentations at regional and national conferences.

ELIGIBILITY:
For Work Packages 1 and 2-

Inclusion Criteria:

1. People diagnosed with Parkinson's or caregiver of someone diagnosed with Parkinson's
2. Able to consent to participate

Exclusion Criteria:

1. Unable to consent to participate

For Work Package 3:

Inclusion Criteria:

1. Have a role in the care of someone with Parkinson's including but not limited to people diagnosed with Parkinson's, caregiver of someone with diagnosed with Parkinson's, healthcare professionals, volunteer sector representative, policy maker or manager
2. Able to consent to participate.

Exclusion criteria:

1. Unable to consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Participants for the interviews will be purposively sampled from Parkinson's clinics in Hampshire and Dorset.
  2. Participants for the national survey will be recruited from Parkinson's clinics in Hampshire and Dorset as well as through Parkinson's UK Research Support Network and Take Part Hub.
  3. Participants for the focus groups will be recruited from Parkinson's clinics in Hampshire and Dorset as well as working with Wessex Parkinson's Excellence Network
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Treatment Burden Experiences | 24 months
  The investigators will describe the key factors that influence participants' experiences of treatment burden
Capacity | 24 months
  The investigators will describe the key factors that influence participants' capacity
Treatment Burden Levels | 24 months
  Treatment burden levels will be measured using the Multimorbidity Treatment Burden Questionnaire (MTBQ):- Overall scores (0-100) categorised as no burden (score 0), low burden (score <10), medium burden (10-22) and high burden (>=22).

SECONDARY OUTCOMES:
Multimorbidity and treatment burden levels | 24 months
  Multimorbidity assessed with self-reported number of co-morbidities
Frailty and treatment burden levels | 24 months
  Frailty assessed using the Program of Research to Integrate Services for the Maintenance of Autonomy (PRISMA-7) screening tool; Score of ≥3 defined as frail
Severity of Parkinson's and treatment burden levels | 24 months
  Severity Parkinson's will be measured using the self-reported Hoehn and Yahr scale (0-5) 0 - No sign of disease
  1. - Unilateral involvement
  2. - Bilateral involvement without impairment of balance
  3. - Mild to moderate bilateral disease; some postural instability; physically independent
  4. - Severe disability; still able to walk or stand unassisted
  5. - Wheelchair bound or bedridden unless aided

CONTACTS AND LOCATIONS:
Overall Officials: Qian Yue Tan, Principal Investigator — University of Southampton
Locations (2):
- United Kingdom (2):
  - Christchurch Hospital, University Hospitals Dorset NHS Foundation Trust, Bournemouth, Dorset
  - Romsey Hospital, Southern Health NHS Foundation Trust, Southampton, Hampshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymised study data will be made available upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The investigators will preserve all study data and keep it available for sharing within the science community for up to 10 years. This timeframe is consistent with the investigators' local university policy.
Access Criteria: Requests for access to anonymised data by other researchers can be submitted by contacting the Principle Investigator. All requests will be carefully considered by the research team.